CLINICAL TRIAL: NCT02416375
Title: A Standardized Multi-centre Analysis of Remote Monitoring in Cystic Fibrosis Adult Patients to Reduce Pulmonary Exacerbations
Brief Title: Home Monitoring to Predict Exacerbation in Cystic Fibrosis
Acronym: SmartCare
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Cystic Fibrosis Trust (Other); King's College Hospital NHS Trust (Other); Royal Brompton & Harefield (Unknown); The Leeds Teaching Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Microsoft Research (Industry); Frimley Park Hospital NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Judy Ryan, Research & Database Manager, Papworth Hospital NHS Foundation Trust
Other Study IDs: PO1955
Record Dates: First submitted 2015-02-10; First posted 2015-04-15 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Daily sputum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Adult Cystic Fibrosis patients

SUMMARY:
The study aims to establish if it is possible for people with Cystic Fibrosis to monitor a number of parameters on a daily basis at home which might predict respiratory infections before they have symptoms and which might also predict treatment failures before this is obvious with conventional measures.

DETAILED DESCRIPTION:
Participants will collect the following clinical information daily: pulse rate and oxygen saturations, wellness and cough scores, spirometry measurements, physical activity, temperature, weight and sleep quantity and quality. The patients will also collect daily sputum samples.

Data will be collected via Bluetooth-enabled devices and transmitted via a Smart-phone to a secure National Health Service approved web-based site to be analyzed.

The information obtained will allow the investigators to develop a software program that will identify signals that can predict the onset of a chest infection before symptoms develop.

The investigators will also measure specific substances in sputum to identify changes before, during and after chest infections. The investigators hope this additional information will enable them to more accurately predict the onset of chest infections in cystic fibrosis.

The results of this study will determine if it is possible to develop a simple sputum test for patients to use at home in combination with other home-based assessments of well-being to provide an early warning system of a chest infection before patients feel unwell.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Cystic Fibrosis based on genetic testing and/or sweat chloride.
2. Age ≥ 18 years of age.
3. A history of at least 1 acute pulmonary exacerbation in the past 12 months.
4. Able to provide written informed consent.
5. Willing and able to produce daily sputum samples.
6. Willing and able to provide daily telemetric measure of several physiological parameters.

Exclusion Criteria:

1. Patients unable to provide written informed consent
2. Patients unable to produce daily sputum samples
3. Less than 1 infective pulmonary exacerbation in 12 months
4. Lung transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Cystic Fibrosis patients who produce sputum daily and have not had a previous organ transplant, with a history of at least one pulmoanry exacerbation within the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Home monitoring possible in adult Cystic Fibrosis patients | 6 months
  This will be measured by the number of patients recruited into the study and the patients compliance / adherence to the study protocol

SECONDARY OUTCOMES:
Whether daily monitoring can provide early warning of a new chest infection | 6 months
  Identification of predictive signals for early detection of an acute pulmonary exacerbations and treatment response in patients with cystic fibrosis
Development of a web-based machine learning tool | 6 months
  Development of a web-based machine learning associated tool to predict acute pulmonary exacerbation and treatment response in patients with cystic fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Floto, Prof, Principal Investigator — Papworth Hospital NHS
Locations (2):
- United Kingdom (2):
  - Papworth Hospital NHS Trust, Cambridge, Cambridgeshire
  - Papworth Hospital NHS Trust, Cambridge